CLINICAL TRIAL: NCT05926817
Title: Effect of Virtual Reality Intervention on Hospitalized Patients With Acute Pain After Thoracoscopic Surgery: A Randomized Clinical Trial
Brief Title: Effect of Virtual Reality on Patients With Acute Pain After Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Weibo Cao, Principal investigator, Tianjin Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB2021-YX-173-01
Record Dates: First submitted 2023-06-14; First posted 2023-07-03 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Virtual Reality; Acute Postoperative Pain; Thoracic Surgery, Video-Assisted
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Postoperative standard analgesia was administered to patients in the control group.
- Placebo-VR group (Placebo Comparator): Patients in the Placebo-VR group watched a 10-minute relaxation-based 2D film through VR headsets along with receiving conventional analgesia.
  Interventions: Device: Placebo-VR headsets
- QTC-VR group (Experimental): Patients in the QTC-VR group engaged in 10-minute interactive pain relief 3D VR programs while wearing VR headsets along with receiving conventional analgesia.
  Interventions: Device: QTC-VR headsets

INTERVENTIONS:
Device: Placebo-VR headsets — Patients in the Placebo-VR group watched a 10-minute relaxation-based 2D film through VR headsets along with receiving conventional analgesia.
  Arms: Placebo-VR group
Device: QTC-VR headsets — Patients in the QTC-VR group engaged in 10-minute interactive pain relief 3D VR programs while wearing VR headsets along with receiving conventional analgesia.
  Arms: QTC-VR group

SUMMARY:
Immersive virtual reality (VR) as a non-pharmaceutical technology may deliver effective behavioral therapies for postsurgical patients with acute pain. To determine the analgesic effects of VR on patients after thoracoscopic surgery. The investigators conducted a randomized clinical trial to determine the postoperative effect of VR on pain relief in patients undergoing thoracoscopic surgery.

DETAILED DESCRIPTION:
Immersive virtual reality (VR) as a non-pharmaceutical technology may deliver effective behavioral therapies for postsurgical patients with acute pain. Patients in the QTC-VR group had to participate in 15-minute interactive games wearing 3D-VR headsets. QTC-VR intervention had functions for breath-relaxation and attention-concentration training. It instructed the patients to breathe deeply with the marine animal's swimming relaxation rhythm and to constantly switch the vision field by rotating their heads and necks to catch animals. Therefore, the investigators conducted a randomized clinical trial to determine the postoperative effect of QTC-VR on pain relief in patients undergoing thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's age is ≥ 18, regardless of gender.
2. Within one day after thoracoscopic surgery.
3. The NRS of postoperative pain is ≥ four.
4. Having specific internet knowledge and mobile phone reading and writing abilities.
5. Patients voluntarily sign the informed consent form and are willing to complete the follow-up according to the trial protocol.

Exclusion Criteria:

1. Patients have severe cognitive disorders.
2. Patients with previous diagnoses of epilepsy, dementia, migraine, or other neurological diseases may have difficulty using the VR headset.
3. Patients are sensitive to light stimulation.
4. Patients are without stereopsis or with severe hearing impairment.
5. Patients with trauma to the eyes, face, or neck are not comfortable using VR headsets.
6. Patients have severe heart, liver, kidney, blood, digestive, and nervous diseases.
7. Patients previously used the VR headset but found it ineffective.
8. Patients have a history of severe alcoholism, long-term heavy drinking, and symptoms of alcohol dependence.
9. Patients have participated in any analgesic intervention study in the past week.
10. Women have pregnancy plans during the follow-up period of the study.
11. Patients and their families work in digital health or pharmaceutical companies for acute or chronic pain management.
12. Patients cannot use electronic devices such as smartphones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Change in Pain intensity evaluating by the numerical rating scale (NRS) | Evaluating pain intensity among postoperative patients 10 minutes prior to and 30 minutes following the intervention
  The primary outcome was the change in pain intensity following the QTC-VR and Placebo-VR intervention.

SECONDARY OUTCOMES:
Pain-related interference on patients' mood by the brief pain inventory (BPI) | The patients' pain interference was evaluated within 30 minutes of the intervention.
  Secondary outcomes included the pain interference on their mood.
Pain-related interference on patients' sleep by the brief pain inventory (BPI) | The patients' pain interference was evaluated within 30 minutes of the intervention.
  Secondary outcomes included the pain interference on their sleep.
Pain-related interference on patients' daily life by the brief pain inventory (BPI) | The patients' pain interference was evaluated within 30 minutes of the intervention.
  Secondary outcomes included the pain interference on their daily life.
Pain-related interference on patients' interest in life by the brief pain inventory (BPI) | The patients' pain interference was evaluated within 30 minutes of the intervention.
  Secondary outcomes included the pain interference on their enjoyment of life.
Pain-related interference on patients' walking ability by the brief pain inventory (BPI) | The patients' pain interference was evaluated within 30 minutes of the intervention.
  Secondary outcomes included the pain interference on their walking ability.
Patient satisfaction regarding the VR by the satisfaction evaluation form | We assessed patient satisfaction with VR after the end of the third day of the VR intervention.
  Secondary outcomes included patient satisfaction regarding the VR intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Song Xu, Study Director — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No